CLINICAL TRIAL: NCT05003804
Title: A Phase 1b/2, Randomized, Double-blind, Placebo-controlled, Multi-center Study of STMC-103H in Neonates and Infants at Risk for Developing Allergic Disease
Brief Title: Allergic Disease Onset Prevention Study
Acronym: adored
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Siolta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STMC-103H-102
Record Dates: First submitted 2021-08-04; First posted 2021-08-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis; Type 1 Hypersensitivity
MeSH Terms: conditions — Dermatitis, Atopic; Hypersensitivity, Immediate

STUDY DESIGN:
Intervention Model Description: Participants will be enrolled in a three-part sequential approach (Parts A1, A2, and B). Part A will enroll at risk participants of 1 year to less than 6 years of age; after safety review, Part A2 will enroll at risk participants of 1 month to less than 12 months of age; and after safety review, Part B will enroll at -risk participants between 0 and 14 days of life.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- STMC-103H Part A1 (Experimental): Once daily dosing with one capsule of STMC-103H mixed with milk, formula, or a milk product for 28 days
  Interventions: Biological: STMC-103H
- Placebo Part A1 (Placebo Comparator): Once daily dosing with one capsule of placebo mixed with milk, formula, or a milk product for 28 days
  Interventions: Biological: Placebo
- STMC-102H Part A2 (Experimental): Once daily dosing with one capsule of STMC-103H mixed with milk, formula, or a milk product for 28 days
  Interventions: Biological: STMC-103H
- Placebo Part A2 (Placebo Comparator): Once daily dosing with one capsule of placebo mixed with milk, formula or a milk product for 28 days
  Interventions: Biological: Placebo
- STMC-103H Part B (Experimental): Once daily dosing with one capsule of STMC-103H mixed with breastmilk, formula or a milk product for 336 days
  Interventions: Biological: STMC-103H
- Placebo Part B (Placebo Comparator): Once daily dosing with one capsule of placebo mixed with breastmilk, formula or a milk product for 336 days
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: STMC-103H — STMC-103H is a live biotherapeutic product (LBP) containing a consortium of intestinal bacteria
  Arms: STMC-102H Part A2; STMC-103H Part A1; STMC-103H Part B
Biological: Placebo — Powder containing excipients found in STMC-103H: magnesium stearate, mannitol and silicon dioxide.
  Arms: Placebo Part A1; Placebo Part A2; Placebo Part B

SUMMARY:
This is a Phase 1b/2, randomized, double-blind, multi-center study to evaluate the safety, tolerability, and preliminary clinical efficacy of STMC-103H in neonates and infants at risk for developing allergic disease (Type 1 hypersensitivity). Subjects will be enrolled in a three-part sequential approach. Participants in the safety-run portion of the study (Part A1: 1 year to <6 years of age and A2: 1 month to <12 months of age) will receive 28 days of treatment with STMC-103H or placebo, followed by 28 days of follow-up. A Data and Safety Monitoring Committee (DSMC) will review safety data after all patients in each part complete 28 days of therapy prior to enrolling the next part. After A2, Part B will enroll 224 patients for 336 days of treatment with STMC-103H or placebo, followed by 336 days of follow-up. Stool, blood, and optional samples will be collected in Parts A2 and part B. Primary safety endpoints are frequency, type and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs), as well as findings on physical exams, vitals, and safety laboratories. The primary efficacy endpoint is incidence of physician-diagnosed atopic dermatitis at day 336.

ELIGIBILITY:
Inclusion Criteria:

* All Parts (A1, A2, B)

  1. Subject's parent(s)/legal representative(s) providing consent must be 18 years or older
  2. Biological mother and/or biological father and/or full sibling(s), have a history of asthma, atopic dermatitis, food allergy, or allergic rhinitis as determined by the screening questionnaire
  3. Subject's parent(s)/legal representative(s) (if appropriate according to local laws) is/are willing and able to give informed consent for participation in the study
  4. Subject's parent(s)/legal representative(s) (if appropriate according to local laws) is/are willing and able, in the PI's opinion, to comply with all study requirements

Part A1 Only

Inclusion criteria 1-4 for all parts plus:

5 (A1). Subject is between 1 year and < 6 years old at the time of enrollment

Part A2 Only

Inclusion criteria 1-4 for all parts plus:

5 (A2). Subject is between 28 days and < 12 months of life at the time of enrollment 6 (A2). Subject's parent(s)/legal representative(s) do not plan to give probiotics (including infant formula that contain probiotics) to the subject during the trial

Part B Only

Inclusion criteria 1-4 for all parts plus:

5 (B). Subject is ≤ 14 days of life at the time of enrollment. Sites should make every effort to enroll newborns as soon as possible after birth.

6 (B). Subject has a birthweight ≥ 2.5 kg and ≤ 4.5 kg 7 (B). Subject's parent(s)/legal representative(s) do not plan to give probiotics (including infant formula that contain probiotics) to the subject from the time of birth to the end of the trial.

Exclusion Criteria:

* All Parts (A1, A2, B)

  1. Subject's twin (or higher order multiple) is enrolled in STMC-103H-102
  2. Subject has any congenital abnormalities or condition, significant disease, illness, physical exam finding, or disorder that, in the opinion of the PI, may put the subject at safety risk or is likely to hinder feeding or affect metabolism that may influence the results of the study. (Neonatal hyperbilirubinemia (jaundice), including jaundice that requires phototherapy, should not be considered exclusionary).
  3. Subject is acutely ill or on systemic antibiotics at the time of enrollment
  4. Subject is participating in another interventional clinical study involving investigational medication, formula, probiotic, or prebiotic use within 30 days (or five half-lives, whichever is longer) of this study
  5. Subject has evidence of immune deficiency/immune compromise in the judgment of the investigator

Part B Only

Exclusion Criteria 1-5 for all parts plus:

6 (B). Subject was born at < 35 weeks' gestation 7 (B). Biological maternal medical condition during the pregnancy that, in the opinion of the PI, may put the subject at risk because of participation in the study. (Maternal antibiotics during the time of delivery should not be considered exclusionary.)

Ages: 0 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 283 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-11-26 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Part A1 and A2: Assess safety and tolerability of STMC-103H in children and infants at risk for development of allergic disease by assessing adverse events (AE), serious adverse events (SAE), and AEs of special interest | Through 56 days of study
  Frequency, type, and severity of AEs and SAEs, including AEs of special interest (AESI) as in Appendix 9 (Adverse Events of Special Interest) and Appendix 10 (Adverse Event Grading Scale)
Part B: Assess the safety, tolerability of STMC-103H in neonate and infants subjects at risk for development of atopic disease by monitoring AEs, SAEs, AESI, physical exam findings, and clinical safety laboratories. | Through 672 days of study
  Frequency, type and severity of AEs, SAEs, and AESIs as in Appendix 9 (Adverse Events of Special Interest) and Appendix 10 (Adverse Event Grading Scale), as well as clinically significant findings on physical examinations including growth (length, weight, height and head circumference) and vital signs (RR, HR, and temperature); clinical safety laboratories including complete blood count with manual differential and blood chemistry
Part B: Primary Efficacy Endpoint: Incidence of physician-diagnosed atopic dermatitis at 336 days | Day 336
  Incidence of physician-diagnosed atopic dermatitis at 336 days in STMC-103H-treated subjects compared to placebo

SECONDARY OUTCOMES:
Part B Secondary Efficacy Endpoint - physician-diagnosed atopic dermatitis | At days 168 and 672
  Incidence of physician-diagnosed atopic dermatitis
Part B - Secondary Efficacy Endpoint - atopic disease assessments | At days 168, 336 and 672
  Proportion of subjects who develop any atopic disease (atopic dermatitis, food allergy, allergic rhinitis/conjunctivitis, asthma)
Part B Secondary Efficacy Endpoint - incidence of sensitization to food and aeroallergen | At days 168, 336, and 672
  Incidence of sensitization to food and aeroallergen as measured by specific serum IgE levels
Part B Secondary Efficacy Endpoint - incidence of food allergy, allergic rhinitis/conjunctivitis, urticaria, and wheezing illness/asthma | At days 168, 336, and 672
  Incidence of physician-diagnosed food allergy, allergic rhinitis/conjunctivitis, urticaria and wheezing illnesses/asthma using physician assessment, Allergic Disease Assessment and Diagnosis questionnaire, and Allergic Disease Diagnostic Criteria & Severity Evaluation
Part B Secondary Efficacy Endpoint - Time to atopic dermatitis diagnosis | Through 672 days of study
  Time to atopic dermatitis diagnosis by physician assessment
Part B Secondary Efficacy Endpoint - Time to first wheezing episode | Through 672 days of study
  Time to first wheezing episode by physician assessment
Part B Secondary Efficacy Endpoint - severity of atopic dermatitis by Investigator Global Assessment x Body Surface Area (IGAxBSA) assessment | At days 168, 336 and 672
  Severity of atopic dermatitis by IGAxBSA assessment
Part B Secondary Efficacy Endpoint - severity of atopic dermatitis by Severity Scoring Of Atopic Dermatitis (SCORAD) assessment | At days 168, 336 and 672
  Severity of atopic dermatitis by SCORAD assessment
Part B Secondary Efficacy Endpoint - Severity of Wheezing Illness/Asthma | At days 68, 336, and 672 days
  Severity of wheezing illness/asthma by Wheezing Severity Assessment
Part B Secondary Efficacy Endpoint - use of concomitant medications for allergic symptoms or diagnosis | Through 672 days of study
  Concomitant medications prescribed/used for allergic symptoms or diagnosis and use of rescue medications for atopic dermatitis and wheezing/asthma
Part B Secondary Efficacy Endpoint - Total Serum IgE | At days 168, 336, and 672
  Total serum IgE levels
Part B Secondary Efficacy Endpoint - Peripheral Eosinophil Counts | At day 336
  Peripheral eosinophil counts by automated differential

OTHER OUTCOMES:
Part B Key Exploratory Endpoint - Mean fecal concentration of 12,13-diHOME | At day 336
  Mean fecal concentration of 12,13-diHOME measured in stool sample in STMC-103H arm as compared to placebo arm

CONTACTS AND LOCATIONS:
Locations (31):
- United States (24):
  - University of Arizona Health Sciences, Tucson, Arizona
  - Arkansas Children's Research Institute, Little Rock, Arkansas
  - UCLA Health, Los Angeles, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Lurie Children's Hospital, Chicago, Illinois
  - University of Chicago Medicine, Chicago, Illinois
  - Riley Children's Health at University of Indiana, Indianapolis, Indiana
  - Johns Hopkins University School of Medicine, Baltimore, MD, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health, Ann Arbor, Michigan
  - Northwell Healthcare, Great Neck, New York
  - NYU Langone Fink Children's, New York, New York
  - Mt. Sinai Jaffe Allergy Institute, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Tribe Clinical Research, Greenville, South Carolina
  - Coastal Pediatrics Research, Summerville, South Carolina
  - Dell Medical School at UT Austin, Austin, Texas
  - UT Southwestern/Children's Health, Dallas, Texas
  - Seattle Allergy and Asthma Research Institute, Seattle, Washington
  - Univ. of Wisconsin-Madison/Jackson Research Group, Madison, Wisconsin
- Australia (6):
  - The Children's Hospital at Westmead, Westmead, New South Wales
  - Queensland Children's Hospital, South Brisbane, Queensland
  - The Women's and Children's Hospital, Adelaide, South Australia
  - Monash Children's Hospital, Clayton, Victoria
  - Murdoch Children's Research Institute, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Centro de Neumologia Pediatrica, Caguas, Puerto Rico, Puerto Rico

IPD SHARING:
Plan to Share IPD: No